CLINICAL TRIAL: NCT03965689
Title: A Phase 2 Study of MLN4924 (Pevonedistat) in Combination With Carboplatin and Paclitaxel in Advanced NSCLC Previously Treated With Immunotherapy
Brief Title: Testing the Combination of MLN4924 (Pevonedistat), Carboplatin, and Paclitaxel in Patients With Advanced Non-small Cell Lung Cancer (NSCLC) Who Have Previously Been Treated With Immunotherapy
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2019-03212; NCI-2019-03212 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); NCI10266; 10266 (Other: JHU Sidney Kimmel Comprehensive Cancer Center LAO); 10266 (Other: CTEP); UM1CA186691 (NIH); UM1CA186716 (NIH)
Record Dates: First submitted 2019-05-27; First posted 2019-05-29 (Actual); Results first posted 2023-12-15 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-09

CONDITIONS: Metastatic Lung Non-Small Cell Squamous Carcinoma; Metastatic Lung Non-Squamous Non-Small Cell Carcinoma; Stage IIIB Lung Cancer AJCC v8; Stage IV Lung Cancer AJCC v8; Stage IVA Lung Cancer AJCC v8; Stage IVB Lung Cancer AJCC v8; Unresectable Lung Non-Small Cell Carcinoma; Unresectable Lung Non-Squamous Non-Small Cell Carcinoma
MeSH Terms: conditions — Lung Neoplasms | interventions — Carboplatin; Paclitaxel; Taxes; pevonedistat

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (paclitaxel, carboplatin, pevonedistat) (Experimental): Patients receive paclitaxel IV over 3 hours on day 1, carboplatin IV over 30-60 minutes on day 1, and pevonedistat IV over 1 hour on days 1, 3, and 5. Treatment repeats every 21 days for at least 4 cycles in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Carboplatin; Drug: Paclitaxel; Drug: Pevonedistat

INTERVENTIONS:
Drug: Carboplatin — Given IV
  Other Names: Blastocarb; Carboplat; Carboplatin Hexal; Carboplatino; Carboplatinum; Carbosin; Carbosol; Carbotec; CBDCA; Displata; Ercar; JM-8; JM8; Nealorin; Novoplatinum; Paraplatin; Paraplatin AQ; Paraplatine; Platinwas; Ribocarbo
Drug: Paclitaxel — Given IV
  Other Names: Anzatax; Asotax; Bristaxol; Praxel; Taxol; Taxol Konzentrat
Drug: Pevonedistat — Given IV
  Other Names: MLN4924; Nedd8-Activating Enzyme Inhibitor MLN4924

SUMMARY:
This phase II trial studies how well MLN4924 (pevonedistat), carboplatin, and paclitaxel work in treating patients with stage IIIB or IV non-small cell lung cancer. Pevonedistat may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth. Chemotherapy drugs, such as carboplatin and paclitaxel, work in different ways to stop the growth of cancer cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Giving pevonedistat together with carboplatin and paclitaxel may work better in treating patients with non-small cell lung cancer when compared with other standard chemotherapy drugs.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To determine the overall response rate (ORR) of patients with advanced non-small cell lung cancer (NSCLC) treated with pevonedistat (MLN4924 [pevonedistat]) in combination with carboplatin and paclitaxel.

SECONDARY OBJECTIVES:

I. To estimate the progression-free survival (PFS) of patients with advanced NSCLC treated with MLN4924 (pevonedistat) in combination with carboplatin and paclitaxel.

II. To estimate the overall survival (OS) of patients with advanced NSCLC treated with MLN4924 (pevonedistat) in combination with carboplatin and paclitaxel.

III. To evaluate the safety profile of MLN4924 (pevonedistat) in combination with carboplatin and paclitaxel.

CORRELATIVE OBJECTIVES:

I. To evaluate expression of nuclear factor-erythroid 2 p45-related factor 2 (NRF2) target genes NAD(P)H: quinone oxidoreductase1 (NQO1) and the cysteine/glutamate antiporter solute carrier family 7 member 11 (SCL7A11).

II. To determine expression of pharmacodynamic markers induced by neural precursor cell expressed developmentally downregulated protein 8 (NEDD-8) activating enzyme (NAE) inhibition: cyclic AMP-dependent transcription factor (ATF3), beta 2 microglobulin (B2M), glutamate-cysteine ligase regulatory subunit (GCLM), glutathione-disulfide reductase (GSR), deoxyribonucleic acid (DNA)-3-methyladenine (MAG1), ribosomal protein lateral stalk subunit P0 (RPLPO), sulfiredoxin-1 (SRXN1), thioredoxin reductase 1 (TXNRD1), and ubiquitin-conjugating enzyme (UBC).

III. To perform qualitative assessment of tumor NAE1 and ubiquitin-conjugating enzyme E2 M (UBC12) protein expression at baseline.

IV. To assess circulating tumor cells (CTCs) for DNA damage repair pathway alterations (i.e., gamma H2AX induction, RAD51).

V. To evaluate pharmacokinetic (PK) parameters of MLN4924 (pevonedistat) when given in combination with paclitaxel and carboplatin.

OUTLINE:

Patients receive paclitaxel intravenously (IV) over 3 hours on day 1, carboplatin IV over 30-60 minutes on day 1, and pevonedistat IV over 1 hour on days 1, 3, and 5. Treatment repeats every 21 days for at least 4 cycles in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, all patients without disease progression are followed up at 30 days, every 3 months for 1 year and then every 6 months until 5 years from end of study treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be >= 18 years old. Because no dosing or adverse event (AE) data are currently available on the use of MLN4924 (pevonedistat) in combination with carboplatin and paclitaxel in patients < 18 years of age, children are excluded from this study, but may be eligible for future pediatric trials.
* Patients must have histologically confirmed stage IIIB or IV NSCLC (squamous or nonsquamous) that is metastatic or unresectable.
* Patients must have measurable disease per Response Evaluation Criteria in Solid Tumors (RECIST) 1.1.
* Patients must have progressed on prior treatment with checkpoint inhibitor (PD-1/PD-L1 inhibitors) either as a single-agent therapy or in combination, as below. Patients will be eligible if there is a contra-indication to checkpoint inhibitor therapy.

  * Patients who have progressed after receiving a checkpoint inhibitor in combination with a platinum-based doublet, as first-line treatment for NSCLC.
  * Patients who have progressed on checkpoint inhibitor as second-line therapy, after receiving a platinum-based doublet as first-line therapy.
  * Patients who have progressed on platinum-based doublet as second-line therapy, after receiving a checkpoint inhibitor as first-line therapy.
* Patients must have disease progression on or after platinum-based chemotherapy for metastatic disease or within 6 months of completion of platinum-based chemotherapy administration as adjuvant/neoadjuvant chemotherapy or concurrent chemoradiation.
* Absolute neutrophil count >= 1,500/mcL.
* Platelet count >= 150,000/mcL.
* Total bilirubin =< 1 x institutional upper limit of normal (ULN). Patients with Gilbert's syndrome may enroll if direct bilirubin =< 1.5 x institutional ULN.
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT]) / alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) =< 3.0 x institutional ULN. Patients with metastatic liver disease may enroll if =< 5 x ULN.
* Glomerular filtration rate (GFR) > 30 mL/min/1.73 m^2.
* Known human immunodeficiency virus (HIV) positive patients who meet the following criteria will be considered eligible:

  * CD4 count > 350 cells/mm^3.
  * Undetectable viral load within the last six months.
  * HIV positive patients must be stable on highly active antiretroviral therapy (HAART). Clinically significant metabolic enzyme inducers are not permitted during this study (e.g., ritonavir, efavirenz, nevirapine).
  * No history of acquired immune deficiency syndrome (AIDS)-defining opportunistic infections.
* Eastern Cooperative Oncology Group (ECOG) performance status 0-1.
* Life expectancy >= 12 weeks.
* Patients are eligible if central nervous system (CNS) metastases are adequately treated and neurological symptoms have returned to baseline or are controlled for at least 2 weeks prior to enrollment. In addition, subjects must be either off corticosteroids, or on stable or decreasing dose of steroids. Patients with leptomeningeal disease are excluded.
* The effects of MLN4924 (pevonedistat) on the developing human fetus are unknown. For this reason and because agents as well as other therapeutic agents used in this trial are known to be teratogenic, women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study or within 4 months of completion, she should inform her treating physician immediately. Men treated or enrolled on this protocol must also agree to use adequate contraception prior to the study, for the duration of study participation, and 4 months after completion of MLN4924 (pevonedistat) administration.

Female patients who:

* Are postmenopausal for at least 1 year before the screening visit, or
* Are surgically sterile, or If they are of childbearing potential,
* Agree to practice 1 highly effective method and 1 additional effective (barrier) method of contraception, at the same time, from the time of signing the informed consent through 4 months after the last dose of study drug (female and male condoms should not be used together), or
* Agree to practice true abstinence, when this is in line with the preferred and usual lifestyle of the subject. (Periodic abstinence [e.g., calendar, ovulation, symptothermal, postovulation methods] withdrawal, spermicides only, and lactational amenorrhea are not acceptable methods of contraception.) Male patients, even if surgically sterilized (i.e., status postvasectomy), who
* Agree to practice effective barrier contraception during the entire study treatment period and through 4 months after the last dose of study drug (female and male condoms should not be used together), OR
* Agree to practice true abstinence, when this is in line with the preferred and usual lifestyle of the subject. (Periodic abstinence [e.g., calendar, ovulation, symptothermal, postovulation methods for the female partner] withdrawal, spermicides only, and lactational amenorrhea are not acceptable methods of contraception.)

  * For patients with evidence of chronic hepatitis B virus (HBV) infection, the HBV viral load must be undetectable on suppressive therapy, if indicated.
  * Patients with a history of hepatitis C virus (HCV) infection must have been treated and cured. For patients with HCV infection who are currently on treatment, they are eligible if they have an undetectable HCV viral load.
  * Patients with a prior or concurrent malignancy whose natural history or treatment does not have the potential to interfere with the safety or efficacy assessment of the investigational regimen are eligible for this trial.
  * Left ventricular ejection fraction (LVEF) >= 50% as assessed by echocardiogram or radionuclide angiography.
  * Ability to understand and the willingness to sign a written informed consent document. Participants with impaired decision-making capacity (IDMC) who have a legally authorized representative (LAR) or caregiver and/or family member available will also be considered eligible.
  * Patients with NSCLC harboring genomic aberrations (e.g. sensitizing EGFR, ALK, ROS1, NTRK, BRAF V600E mutation positive) must have received prior treatment with Food and Drug Administration (FDA) approved targeted therapy for patients for which FDA approved targeted therapies is available.

Exclusion Criteria:

* Patients who have not recovered from AEs due to prior anti-cancer therapy (i.e., have residual toxicities > grade 1) with the exception of alopecia and neuropathy.
* Patients who are receiving any other investigational agents.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to MLN4924 (pevonedistat), carboplatin, or paclitaxel.
* Patients who have had chemotherapy or radiotherapy within 2 weeks (6 weeks for nitrosoureas or mitomycin C) prior to entering the study.
* Patients with uncontrolled intercurrent illness.
* Patients with psychiatric illness/social situations that would limit compliance with study requirements.
* Pregnant women are excluded from this study because MLN4924 (pevonedistat), carboplatin, and paclitaxel have the potential for teratogenic or abortifacient effects. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with MLN4924 (pevonedistat), breastfeeding must be discontinued if the mother is treated with MLN4924 (pevonedistat). These potential risks may also apply to other agents used in this study.
* Female patients who intend to donate eggs (ova) during the course of this study or 4 months after receiving their last dose of study drug(s).
* Male patients who intend to donate sperm during the course of this study or 4 months after receiving their last dose of study drug(s).
* Known cardiopulmonary disease defined as:

  * Unstable angina;
  * Congestive heart failure (New York Heart Association [NYHA] class III or IV;);
  * Myocardial infarction within 6 months prior to first dose (patients who had ischemic heart disease such as acute coronary syndrome [ACS], myocardial infarction, and/or revascularization greater than 6 months before screening and who are without cardiac symptoms may enroll);
  * Symptomatic cardiomyopathy;
  * Clinically significant arrhythmia:

    * History of polymorphic ventricular fibrillation or torsade de pointes,
    * Permanent atrial fibrillation, defined as continuous atrial fibrillation for >= 6 months,
    * Persistent atrial fibrillation, defined as sustained atrial fibrillation lasting > 7 days and/or requiring cardioversion in the 4 weeks before screening,
    * Grade 3 atrial fibrillation defined as symptomatic and incompletely controlled medically, or controlled with device (e.g., pacemaker), or ablation in the past 6 months and
    * Patients with paroxysmal atrial fibrillation or grade < 3 atrial fibrillation for period of at least 6 months are permitted to enroll provided that their rate is controlled on a stable regimen.
  * Clinically symptomatic pulmonary hypertension requiring pharmacologic therapy.
* Peripheral neuropathy that is grade >= 3, or grade 2 with pain on clinical examination during the screening period.
* Uncontrolled high blood pressure (i.e., systolic blood pressure > 180 mmHg, diastolic blood pressure > 95 mmHg).
* Prolonged rate corrected QT (QTc) interval >= 500 msec, calculated according to institutional guidelines.
* Known moderate to severe chronic obstructive pulmonary disease, interstitial lung disease, and pulmonary fibrosis.
* Major surgery within 14 days before the first dose of any study drug or a scheduled surgery during study period.
* Life-threatening illness unrelated to cancer.
* Patients with uncontrolled coagulopathy or bleeding disorder.
* Known hepatic cirrhosis or severe pre-existing hepatic impairment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2020-04-16 (Actual); Primary Completion 2022-09-07 (Actual); Study Completion 2026-03-18 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Ticiana A Leal, Principal Investigator — JHU Sidney Kimmel Comprehensive Cancer Center LAO
Locations (10):
- United States (10):
  - Los Angeles General Medical Center, Los Angeles, California
  - USC / Norris Comprehensive Cancer Center, Los Angeles, California
  - USC Norris Oncology/Hematology-Newport Beach, Newport Beach, California
  - MedStar Georgetown University Hospital, Washington D.C., District of Columbia
  - Moffitt Cancer Center-International Plaza, Tampa, Florida
  - Moffitt Cancer Center - McKinley Campus, Tampa, Florida
  - Moffitt Cancer Center, Tampa, Florida
  - Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - University of Wisconsin Carbone Cancer Center - University Hospital, Madison, Wisconsin

IPD SHARING:
Plan to Share IPD: Yes
NCI is committed to sharing data in accordance with NIH policy. For more details on how clinical trial data is shared, access the link to the NIH data sharing policy page.
URL: https://grants.nih.gov/policy/sharing.htm

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Treatment (Paclitaxel, Carboplatin, Pevonedistat)
Started | 27
Completed | 25
Not Completed | 2
Not completed — Too sick to get study intervention | 2

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (Paclitaxel, Carboplatin, Pevonedistat)
Number analyzed (Participants) | 27
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 15
  >=65 years | 12
Age, Continuous [Median (Full Range); unit: years] | 64 [27 to 77]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12
  Male | 15
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 25
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 6
  White | 19
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 27
Height [Median (Full Range); unit: centimeter (cm)] | 166.5 [146.0 to 189.3]
Weight [Median (Full Range); unit: kilogram (kg)] | 71.8 [44.1 to 134.5]
Body Surface Area (BSA) [Median (Full Range); unit: meters squared (m^2)] | 1.81 [1.41 to 2.66]
Disease Stage [Count of Participants; unit: Participants]
  Advanced Disease (Stage IIIB) | 2
  Metastatic Disease (Stage IV) | 25
Smoking Status [Count of Participants; unit: Participants]
  Current Smoker | 3
  Former Smoker | 19
  Never Smoked | 5

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With an Overall Response
Description: Response will be evaluated at the time all participants completed treatment and using the new international criteria proposed by the revised Response Evaluation Criteria in Solid Tumors (RECIST) guideline (version 1.1). Changes in the largest diameter (unidimensional measurement) of the tumor lesions and the shortest diameter in the case of malignant lymph nodes are used in the RECIST criteria. Patients will be re-evaluated for response every 6 weeks. Overall response is the best response achieved during the study. Complete response (CR) is the disappearance of all lesions; Partial response (PR) is a >= 30% decrease in the sum of the target lesions; Progressive disease (PD) is a >= 20% increase in the sum of the lesions; Stable disease (SD) is between a 20 % increase and 30% decrease in the sum of the lesions.
Time Frame: Up to 2.5 years
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Paclitaxel, Carboplatin, Pevonedistat)
Number analyzed (Participants) | 25
Participants
  Complete Response (CR) | 0
  Partial Response (PR) | 4
  Stable Disease (SD) | 15
  Progressive Disease (PD) | 4
  Not Assessed (NA) | 2

2. Secondary Outcome: Duration of Progression Free Survival (PFS)
Description: Progression free survival (PFS) is defined at the time all participants completed treatment and using Response Evaluation Criteria in Solid Tumors (RECIST v1.1) as >= 20% increase in the sum of target lesions, a measurable increase in a non-target lesion, or the appearance of a new lesion. The duration is measured from the start of treatment to the time of progression or death, whichever occurs first.
Time Frame: Up to 2.5 years
Measure: Median (Full Range); unit: months
Arm/Group | Treatment (Paclitaxel, Carboplatin, Pevonedistat)
Number analyzed (Participants) | 25
months | 3.68 [0.46 to 19.67]

3. Secondary Outcome: Overall Survival (OS)
Description: Defined as the duration of time from start of treatment to time of death or last known date alive at the time all participants completed treatment.
Time Frame: Up to 2.5 years
Measure: Median (Full Range); unit: months
Arm/Group | Treatment (Paclitaxel, Carboplatin, Pevonedistat)
Number analyzed (Participants) | 25
months | 7.73 [0.79 to 21.71]

4. Secondary Outcome: Number of Participants Reporting Grade 3, 4, and 5 Adverse Events
Description: Evaluated by the revised National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 5.0.
Time Frame: 1 year, on average
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Paclitaxel, Carboplatin, Pevonedistat)
Number analyzed (Participants) | 25
Participants
  Grades 3, 4, and 5 | 21
  Grades 1 and 2 | 4

5. Other Pre Specified Outcome: NQO1 Expression Levels
Description: Summarized using descriptive statistics. Ratios of the day 1 pre-treatment over the 6 hours post-infusion levels will be calculated and reported along with the corresponding 95% confidence intervals. A one sample t-test or Wilcoxon Signed Rank test will be used to evaluate changes from the day 1 pre-treatment to the 6 hours post-infusion assessment. A two-sample t-test or nonparametric Wilcoxon Rank Sum test will be used to compared changes in NQO1 expression levels from day 1 pre-treatment to 6 hours post-infusion between responders and non-responders.
Time Frame: Day 1 pre-treatment and 6 hours post-infusion
Reporting Status: Not Posted

6. Other Pre Specified Outcome: SLC7A11 Expression Levels
Description: Summarized using descriptive statistics. Ratios of the day 1 pre-treatment over the 6 hours post-infusion levels will be calculated and reported along with the corresponding 95% confidence intervals. A one sample t-test or Wilcoxon Signed Rank test will be used to evaluate changes from the day 1 pre-treatment to the 6 hours post-infusion assessment. A two-sample t-test or nonparametric Wilcoxon Rank Sum test will be used to compared changes in SLC7A11 expression levels from day 1 pre-treatment to 6 hours post-infusion between responders and non-responders.
Time Frame: Day 1 pre-treatment and 6 hours post-infusion
Reporting Status: Not Posted

7. Other Pre Specified Outcome: NAE1 Expression Levels
Description: Qualitative assessment of tumor NAE1 expression will be conducted by evaluating descriptive summaries of NAE1 expression levels. Changes from the pre-treatment to post-infusion assessment will be evaluated using a paired t-test or nonparametric Wilcoxon Signed Rank test.
Time Frame: Pre-treatment and 6 hours post-infusion on cycle 1, day 1
Reporting Status: Not Posted

8. Other Pre Specified Outcome: UBC12 Expression Level
Description: Qualitative assessment of tumor UBC12 expression will be conducted by evaluating descriptive summaries of UBC12 expression levels. Changes from the pre-treatment to post-infusion assessment will be evaluated using a paired t-test or nonparametric Wilcoxon Signed Rank test.
Time Frame: Pre-treatment and 6 hours post-infusion on cycle 1, day 1
Reporting Status: Not Posted

9. Other Pre Specified Outcome: RAD51 in CTCs
Description: A linear mixed effects model with patient -specific random effects will be utilized to compared changes in RAD51. Changes from the pre-treatment to post-infusion assessment will be evaluated using a paired t-test or nonparametric Wilcoxon Signed Rank test.
Time Frame: Baseline and after treatment with pevonedistat
Reporting Status: Not Posted

10. Other Pre Specified Outcome: GammaH2AX in Circulating Tumor Cells (CTCs)
Description: A linear mixed effects model with patient -specific random effects will be utilized to compared changes in gammaH2AX. Changes from the pre-treatment to post-infusion assessment will be evaluated using a paired t-test or nonparametric Wilcoxon Signed Rank test.
Time Frame: Baseline and after treatment with pevonedistat
Reporting Status: Not Posted

11. Other Pre Specified Outcome: ATF3 Expression Levels
Description: Summarized in terms of means, standard deviations, and ranges, stratified by assessment time point. Changes from the pre-treatment to post-infusion assessment will be evaluated using a paired t-test or nonparametric Wilcoxon Signed Rank test.
Time Frame: Pre-treatment and 6 hours post-infusion on cycle 1, day 1
Reporting Status: Not Posted

12. Other Pre Specified Outcome: B2M Expression Levels
Description: as for outcome 11
Time Frame: Pre-treatment and 6 hours post-infusion on cycle 1, day 1
Reporting Status: Not Posted

13. Other Pre Specified Outcome: GCLM Expression Levels
Description: as for outcome 11
Time Frame: Pre-treatment and 6 hours post-infusion on cycle 1, day 1
Reporting Status: Not Posted

14. Other Pre Specified Outcome: GSR Expression Levels
Description: as for outcome 11
Time Frame: Pre-treatment and 6 hours post-infusion on cycle 1, day 1
Reporting Status: Not Posted

15. Other Pre Specified Outcome: MAG1 Expression Levels
Description: as for outcome 11
Time Frame: Pre-treatment and 6 hours post-infusion on cycle 1, day 1
Reporting Status: Not Posted

16. Other Pre Specified Outcome: RPLP0 Expression Levels
Description: as for outcome 11
Time Frame: Pre-treatment and 6 hours post-infusion on cycle 1, day 1
Reporting Status: Not Posted

17. Other Pre Specified Outcome: SRXN1 Expression Levels
Description: as for outcome 11
Time Frame: Pre-treatment and 6 hours post-infusion on cycle 1, day 1
Reporting Status: Not Posted

18. Other Pre Specified Outcome: TXNRD1 Expression Levels
Description: as for outcome 11
Time Frame: Pre-treatment and 6 hours post-infusion on cycle 1, day 1
Reporting Status: Not Posted

19. Other Pre Specified Outcome: UBC Expression Levels
Description: as for outcome 11
Time Frame: Pre-treatment and 6 hours post-infusion on cycle 1, day 1
Reporting Status: Not Posted

20. Other Pre Specified Outcome: Pharmacokinetics (PK) Parameters
Description: Summarized in terms of means, standard deviations, medians, and ranges, stratified by assessment time point. Changes in PK parameters between assessment time points will be evaluated using a paired t-test.
Time Frame: Pre-treatment and 6 hours post-infusion on cycle 1, day 1
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: From initiation of study therapy to completion of adverse event (AE) observation period. The longest duration for all participants was about 1.75 years.
Arm/Group | Treatment (Paclitaxel, Carboplatin, Pevonedistat)
All-Cause Mortality (participants affected / at risk) | 21/25
Serious Adverse Events (participants affected / at risk) | 16/25
Other Adverse Events (participants affected / at risk) | 25/25
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment (Paclitaxel, Carboplatin, Pevonedistat) (N=25)
Febrile neutropenia (Blood and lymphatic system disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 1
Diverticultis (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Death NOS (General disorders) | 1
Fever (General disorders) | 1
Polytrauma related to motor vehicle accident (General disorders) | 1
Non-cardiac chest pain (General disorders) | 2
COVID-19 Infection (Infections and infestations) | 1
Lung infection (Infections and infestations) | 1
Sepsis (Infections and infestations) | 1
Infusion related reaction (Injury, poisoning and procedural complications) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 2
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 2
Ataxia (Nervous system disorders) | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2
Thromboembolic event (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment (Paclitaxel, Carboplatin, Pevonedistat) (N=25)
Anemia (Blood and lymphatic system disorders) | 15
Sinus bradycardia (Cardiac disorders) | 2
Tachycardia (Cardiac disorders) | 2
Abdominal pain (Gastrointestinal disorders) | 2
Constipation (Gastrointestinal disorders) | 8
Diarrhea (Gastrointestinal disorders) | 4
Nausea (Gastrointestinal disorders) | 11
Vomiting (Gastrointestinal disorders) | 3
Edema limbs (General disorders) | 3
Fatigue (General disorders) | 11
Flu like symptoms (General disorders) | 2
Pain (General disorders) | 6
Papulopustular rash (Infections and infestations) | 2
Transaminitis (Infections and infestations) | 2
Infusion related reaction (Injury, poisoning and procedural complications) | 2
Alanine aminotransferase increased (Investigations) | 15
Alkaline phosphatase increased (Investigations) | 8
Aspartate aminotransferase increased (Investigations) | 15
Blood lactate dehydrogenase increased (Investigations) | 2
Creatinine increased (Investigations) | 4
Lymphocyte count decreased (Investigations) | 5
Neutrophil count decreased (Investigations) | 14
Platelet count decreased (Investigations) | 12
White blood cell decreased (Investigations) | 13
Anorexia (Metabolism and nutrition disorders) | 2
Hyperglycemia (Metabolism and nutrition disorders) | 6
Hyperkalemia (Metabolism and nutrition disorders) | 4
Hyperuricemia (Metabolism and nutrition disorders) | 2
Hypoalbuminemia (Metabolism and nutrition disorders) | 5
Hypocalcemia (Metabolism and nutrition disorders) | 5
Hypokalemia (Metabolism and nutrition disorders) | 7
Hypomagnesemia (Metabolism and nutrition disorders) | 4
Hyponatremia (Metabolism and nutrition disorders) | 5
Hypophosphatemia (Metabolism and nutrition disorders) | 7
Arthralgia (Musculoskeletal and connective tissue disorders) | 4
Chest wall pain (Musculoskeletal and connective tissue disorders) | 2
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 3
Muscle cramp (Musculoskeletal and connective tissue disorders) | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 5
Dizziness (Nervous system disorders) | 5
Paresthesia (Nervous system disorders) | 2
Peripheral sensory neuropathy (Nervous system disorders) | 4
Anxiety (Psychiatric disorders) | 3
Confusion (Psychiatric disorders) | 2
Insomnia (Psychiatric disorders) | 5
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 4
Alopecia (Skin and subcutaneous tissue disorders) | 12
Erythema multiforme (Skin and subcutaneous tissue disorders) | 2
Pruritus (Skin and subcutaneous tissue disorders) | 5
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 4
Hypertension (Vascular disorders) | 3
Hypotension (Vascular disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-12-20): https://cdn.clinicaltrials.gov/large-docs/89/NCT03965689/Prot_SAP_000.pdf
  • Informed Consent Form (2021-12-20): https://cdn.clinicaltrials.gov/large-docs/89/NCT03965689/ICF_001.pdf